CLINICAL TRIAL: NCT06120413
Title: Clinical Evaluation of 18F-LN1 PET/CT for Imaging of Nectin-4 in Urothelial Carcinomas
Brief Title: 18F-LN1 PET/CT in Urothelial Carcinomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Wang, Associate senior physician, Sichuan Provincial People's Hospital
Other Study IDs: SichuanPPH-UCs
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The clinical feasibility of 18F-LN1 PET/CT will be evaluated in 30 patients with urothelial carcinoma, and the results will be compared with those of 18F-FDG.

DETAILED DESCRIPTION:
This study aims to evaluate the recognition efficiency of 18F-LN1 and 18F-FDG PET imaging for tumor target Nectin-4 in patients with urothelial carcinoma. The main method is to compare the results of visually interpreted PET images with histopathological results (through surgery or biopsy), which are the gold standard for final diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* No gender difference
* Patients who have been diagnosed with, or are clinically highly suspected of, urothelial carcinomas and have had no other treatment within 3 months

Exclusion Criteria:

* Hypertension that is difficult to control with medication, and systolic blood pressure exceeding 160mmHg
* Complicated with chronic liver disease, myocardial infarction, stroke
* Female patients who are pregnant (or attempting to become pregnant within six months), breastfeeding, or unwilling to use contraception
* Abnormal cardiopulmonary function or mental state, unable to tolerate prone lying for 20 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically suspected or diagnosed urothelial carcinomas
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of 18F-LN1 and 18F-FDG Uptake in Patients with urothelial carcinoma | 1 mouth
  The correlation between the results of PET images and histopathological results

CONTACTS AND LOCATIONS:
Overall Officials: Hao Wang, Study Director — Sichuan Provincial People's Hospital
Locations (1):
- Departments of Nuclear Medicine, Sichuan Provincial People's Hospital, Chengdu, Sichuan, China